CLINICAL TRIAL: NCT05639556
Title: Strength and Muscle Related Outcomes for Nutrition and Lung Function in CF
Status: Recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: STRONG-CF
Record Dates: First submitted 2022-11-14; First posted 2022-12-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Body Mass Index; Hand Strength; Walk Test; Surveys and Questionnaires; Continuous Glucose Monitoring; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine and stool samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Forced expiratory volume in 1 second (FEV1) <70% predicted during the 12 months prior to enrollment (>50% of measurements, eliminating periods of exacerbation). If no stable spirometry data are available in the 12 months prior to enrollment, from the prior 24 months will be used.
  Interventions: Diagnostic Test: BMI and lean mass index from DXA; Diagnostic Test: Anthropometric Measurements; Diagnostic Test: Hand-grip strength; Diagnostic Test: Six-minute walk Test; Diagnostic Test: Sit-to-Stand Test; Diagnostic Test: Short physical performance battery (SPPB); Diagnostic Test: BIA Sub-study; Diagnostic Test: Accelerometry to assess physical activity; Other: Gastrointestinal (GI) and nutrition questionnaires:; Other: Psychosocial questionnaire: PHQ-8; Other: Psychosocial questionnaire: GAD-7; Other: Psychosocial questionnaire: The Treatment Self-Regulation Questionnaire (TSRQ); Other: Psychosocial questionnaire: CF Fatalism Scale; Other: Psychosocial questionnaire: Body Esteem Scale for Adolescents and Adults (BESAA); Other: 12-month Questionnaire; Other: Oral glucose tolerance testing (OGTT); Device: Continuous glucose monitoring (CGM); Diagnostic Test: Chest CT scans (When available within the past 6 months in medical records); Diagnostic Test: Hologic Dual X-Ray Absorptiometry (DXA); Diagnostic Test: Ultrasound Sub-study of assessment of appendage muscles using ultrasound; Diagnostic Test: Psychosocial questionnaire: Hunger Vital Sign questionnaire; Other: Respiratory symptom questionnaire: CRISS; Diagnostic Test: Spirometry; Other: Psychosocial questionnaire: Additional Health Questionnaire; Other: CF Management Questionnaire; Other: Food Frequency Questionnaire
- Cohort 2: FEV1 ≥70% predicted during the 12 months prior to enrollment (>50% of measurements, eliminating periods of exacerbation).
  Interventions: Diagnostic Test: BMI and lean mass index from DXA; Diagnostic Test: Anthropometric Measurements; Diagnostic Test: Hand-grip strength; Diagnostic Test: Six-minute walk Test; Diagnostic Test: Sit-to-Stand Test; Diagnostic Test: Short physical performance battery (SPPB); Diagnostic Test: BIA Sub-study; Diagnostic Test: Accelerometry to assess physical activity; Other: Gastrointestinal (GI) and nutrition questionnaires:; Other: Psychosocial questionnaire: PHQ-8; Other: Psychosocial questionnaire: GAD-7; Other: Psychosocial questionnaire: The Treatment Self-Regulation Questionnaire (TSRQ); Other: Psychosocial questionnaire: CF Fatalism Scale; Other: Psychosocial questionnaire: Body Esteem Scale for Adolescents and Adults (BESAA); Other: 12-month Questionnaire; Other: Oral glucose tolerance testing (OGTT); Device: Continuous glucose monitoring (CGM); Diagnostic Test: Chest CT scans (When available within the past 6 months in medical records); Diagnostic Test: Hologic Dual X-Ray Absorptiometry (DXA); Diagnostic Test: Ultrasound Sub-study of assessment of appendage muscles using ultrasound; Diagnostic Test: Psychosocial questionnaire: Hunger Vital Sign questionnaire; Other: Respiratory symptom questionnaire: CRISS; Diagnostic Test: Spirometry; Other: Psychosocial questionnaire: Additional Health Questionnaire; Other: CF Management Questionnaire; Other: Food Frequency Questionnaire

INTERVENTIONS:
Diagnostic Test: BMI and lean mass index from DXA — Estimate and compare correlation between lean mass index from DXA and BMI
Diagnostic Test: Anthropometric Measurements — Skinfold will be assessed with calipers. Circumference will be measured with a tape measure.
Diagnostic Test: Hand-grip strength — A small, handheld dynamometer will be used to measure grip strength, a measure of function, on each hand.
Diagnostic Test: Six-minute walk Test — This will be another functional assessment of fitness. Participants will be asked to walk at their normal pace for 6 minutes.The total distance walked in that time will be measured.
Diagnostic Test: Sit-to-Stand Test — This will be used as a functional assessment of fitness and lower extremity strength. Participants will start seated on a chair and be asked to complete as many sit-to-stand repetitions without using their arms for one minute.
Diagnostic Test: Short physical performance battery (SPPB) — This is an assessment of frailty. The test is completed in approximately 8 minutes. The test consists of 3 assessments: 1) Balance tests where the participant stands and tries to balance with their feet in various positions for 10 seconds each without assistance (side-by-side, heel-to-side, and heel-to-toe); 2) Two 4-meter gait speed tests; and 3) Chair-stand tests (single chair stand, 5 chair stands).
Diagnostic Test: BIA Sub-study — A minimum of 50 individuals will be enrolled. Body composition will be assessed at each study visit using study bioelectrical impendence analysis (BIA).
Diagnostic Test: Accelerometry to assess physical activity — Participants will be provided with a wrist-worn accelerometer/heart rate monitor at the baseline study visit and asked to wear it continuously for at least 3-10 days (two weekdays, one weekend day). Approximately every 3 months, the participant will be asked to again wear the accelerometer. Participants will be able to keep their accelerometers.
Other: Gastrointestinal (GI) and nutrition questionnaires: — Subjects will complete surveys regarding gastrointestinal (GI) symptoms, including the Patient Assessment of Constipation (PAC-SYM) Score, Patient Assessment of Gastrointestinal Symptoms (PACGI-SYM) Score, the Bristol Stool Chart, and the scored Patient-Generated Subjective Global Assessment (PG-SGA).
Other: Psychosocial questionnaire: PHQ-8 — This is an 8-item scale that measures depressive symptoms over the past two weeks.
Other: Psychosocial questionnaire: GAD-7 — This is a 7-items scale that measures anxiety symptoms over the past two weeks, from not at all to nearly every day.
Other: Psychosocial questionnaire: The Treatment Self-Regulation Questionnaire (TSRQ) — This is a 15-item scale that assesses the degree to which participants' motivation is autonomous or self-regulated.
Other: Psychosocial questionnaire: CF Fatalism Scale — The CF Fatalism Scale measures the belief in a lack of personal power or control over one's future and has 13 items.
Other: Psychosocial questionnaire: Body Esteem Scale for Adolescents and Adults (BESAA) — The Body Esteem Scale for Adolescents and Adults (BESAA) is 23-item measurement of self-evaluations of one's body or appearance.
Other: 12-month Questionnaire — A short questionnaire designed to explore participants' perspectives of the acceptability and feasibility of nutritional assessments used in STRONG-CF will be given to all study participants at the end of the study.
Other: Oral glucose tolerance testing (OGTT) — For subjects without previously diagnosed CFRD, an OGTT will be performed at baseline and 12-months with samples analyzed at the central lab.
Device: Continuous glucose monitoring (CGM) — Subjects will wear a Dexcom G6Pro sensor in blinded mode for three 10-day periods to collect comprehensive glucose data.
Diagnostic Test: Chest CT scans (When available within the past 6 months in medical records) — Standard of Care chest CT images will be drawn from the medical record, as available, from enrolled participants. FEV1 measurements prior to chest CT scans will be recorded to account for possible illness occurring at the time of scanning. Quantitative assessment of the pectoralis muscle area will be performed on the first single axial image above the aortic arch. Any additional standard of care chest CT's that are performed while the participant is enrolled in the study will also be collected and have a quantitative assessment of the pectoralis muscle performed.
Diagnostic Test: Hologic Dual X-Ray Absorptiometry (DXA) — DXA measurements for whole body, total hip and lumbar spine will be acquired using the Hologic DXA and standard positioning as noted in the DXA Manual of Operations. DXA will be used to estimate total and regional body composition, which will include body fat and lean body mass. This will be used as the gold standard from which to validate BIA and MAMC.
Diagnostic Test: Ultrasound Sub-study of assessment of appendage muscles using ultrasound — A minimum of 50 individuals will be enrolled. At each study visit, participants will undergo ultrasound muscle measurements (cross-sectional area and muscle thickness) of the biceps and quadriceps on each (left and right) side of the body (4 total areas). These measurements will be obtained in triplicate for each patient.
Diagnostic Test: Psychosocial questionnaire: Hunger Vital Sign questionnaire — Screening tool for identifying households at risk of food insecurity and poor health outcomes linked to food insecurity with 3-items over the last 12 months.
Other: Respiratory symptom questionnaire: CRISS — Chronic Respiratory Infection Symptom Score (CRISS) is an 8-item respiratory symptom questionnaire covering the last 24-hours.
Diagnostic Test: Spirometry — Spirometry will be performed in accordance with the current American Thoracic Society recommendations for the performance and interpretation of tests.
Other: Psychosocial questionnaire: Additional Health Questionnaire — Single question over the last 3 months/90 days about cannabis use for GI problems and appetite. The clinical sites will not see the responses to this question. It will be completed by the participant online either during the study visit or at home.
Other: CF Management Questionnaire — Assessment of prior 12-month management of cystic fibrosis, including treatments, medication intake and hospitalizations. This questionnaire will only be completed at 24- and 36- month visits.
Other: Food Frequency Questionnaire — Assessment of prior 12-month nutritional intake being completed at Baseline (no later than 6-month visit) and 12-month visit.

SUMMARY:
The goal of the study is to examine multiple markers of anthropometrics, body composition, sarcopenia and frailty and compare them to dual energy X-ray absorptiometry (DXA) output, which is considered the current clinical gold-standard tool to measure body composition. The result of this study will provide detailed data regarding the nutrition and body composition within this Cystic Fibrosis population and also provide a baseline evaluation for use of these biomarkers in the future studies including evaluation of nutritional intervention. Further, the study will also include psychosocial and other patient-reported outcomes and medical contributors to understand their contributions to the nutritional failure in the adult advanced lung disease population. Finally, the study will evaluate both established and emerging nutritional and body composition parameters and link them to clinical outcomes in adults with CF across the spectrum of pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Participants are eligible if their percentage of predicated forced expiratory volume in 1 second (ppFEV1) is <70% during the 12 months prior to enrollment (>50% of measurements, eliminating periods of exacerbation)
* Cohort 2: Participants are eligible if their percentage of predicted forced expiratory volume in 1 second (ppFEV1) is 70% or greater during the 12 months prior to enrollment (>50% of measurements, eliminating periods of exacerbation).
* Both cohorts match by age, gender, race and CFTR genotype severity.

Exclusion Criteria:

* No prior solid organ transplantation
* No initiation of an investigation drug within 28 days prior to and including Baseline Visit.
* No initiation of new chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, Cayston, CFTR modulator, etc.) within 28 days prior to and including Baseline visit.
* No acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within 14 days prior to and including Baseline visit.
* For the BIA sub-study - Individuals with an implanted pacemaker will be excluded.
* No initiation of a drug for weight loss (such as a GLP-1 receptor agonist) or bariatric surgery within 6-months prior to and including the Baseline visit.
* Patients with continued rapid change or extreme GI symptoms related to weight loss therapy should be excluded at the discretion of the study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults 18 and older with a confirmed diagnostic of cystic fibrosis, identified genotypes (when available), no prior solid organ transplant, and not pregnant or planning on becoming pregnant during the 1st year of the study. Participants receiving a lung transplantation while enrolled in the study will not need to be withdrawn.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between DXA lean mass index and BMI | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and BMI (kg/m2)
Correlation between DXA lean mass index and mid-arm muscle circumference | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and mid-arm muscle circumference (cm)
Correlation between DXA lean mass index and hand-grip strength | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and hand-grip strength (kg)
Correlation between DXA lean mass index and the 6-minute walk distance traveled | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and 6-minute walk (distance traveled in six minutes)
Correlation between DXA lean mass index and the 1-minute sit-to-stand number of repetitions | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and 1-minute sit-to-stand (number of sit-to-stand repetitions in one minute)
Correlation between DXA lean mass index and Short Physical Performance Battery frailty score | Baseline and 1 year
  Estimate and compare correlation between lean mass index from DXA (kg/m2) and Short Physical Performance Battery frailty score (total points)

SECONDARY OUTCOMES:
Characterize lean mass index from DXA cross-sectionally and longitudinally | Baseline and 1 year
  Characterize lean mass index from DXA cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize BMI cross-sectionally and longitudinally | Baseline and 1 year
  Characterize lean mass index from BMI cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize mid-arm measurement circumference cross-sectionally and longitudinally | Baseline and 1 year
  Characterize lean mass index from mid-arm circumference measurements cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize hand-grip strength cross-sectionally and longitudinally | Baseline and 1 year
  Characterize hand-grip strength cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize 1 minute sit-to-stand repetitions cross-sectionally and longitudinally | Baseline and 1 year
  Characterize the 1 minute sit-to-stand repetitions cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize mid-arm 6-minute walk test distance traveled cross-sectionally and longitudinally | Baseline and 1 year
  Characterize the 6-minute walk test distance traveled cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Characterize the Short Physical Performance Battery frailty score cross-sectionally and longitudinally | Baseline and 1 year
  Characterize the Short Physical Performance Battery frailty score cross-sectionally (at enrollment) and longitudinally (post-enrollment changes) based on descriptive statistics and evaluate variance
Compare lean mass index from DXA between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare lean mass index from DXA between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare BMI between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare BMI between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare lean mass index from mid-arm muscle circumference between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare lean mass index from mid-arm muscle circumference between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare hand-grip strength between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare hand-grip strength between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare the 1-minute sit-to-stand repetitions between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare the 1-minute sit-to-stand repetitions between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare the 6-minute walk test distance between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare the 6-minute walk test distance between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Compare the Short Physical Performance Battery frailty score between participants with FEV1 <70% to matched participants with FEV1 ≥70% | Baseline and 1 year
  Compare the Short Physical Performance Battery frailty score between participants with FEV1 <70% to matched participants with FEV1 ≥70%.
Evaluate mean glucose in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate mean glucose from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate % time above 140 mg/dL in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate % time above 140 mg/dL from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate % time above 180 mg/dL in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate % time above 180 mg/dL from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate peak glucose in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate peak glucose from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate % time below 70 mg/dL in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate % time below 70 mg/dL from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate % time below 54 mg/dL in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate % time below 54 mg/dL from continuous glucose measurement data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate the standard deviation in CGM glucose data in participants with FEV1 <70% and matched participants with FEV1 ≥70% | Baseline and 1 year
  Evaluate the standard deviation in CGM glucose data in participants with FEV1 <70% and matched participants with FEV1 ≥70%
Evaluate the coefficient of variation in CGM glucose data in participants with FEV1 <70% and matched participants with FEV1 ≥70% participants | Baseline and 1 year
  Evaluate the coefficient of variation in CGM glucose data in participants with FEV1 <70% and matched participants with FEV1 ≥70% participants

CONTACTS AND LOCATIONS:
Overall Officials: Adam Stein, Principal Investigator — Northwestern University; Jessica Alvarez, Principal Investigator — Emory University; Melissa Putman, Principal Investigator — Massachusetts General Hospital
Locations (24):
- United States (24):
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Boston Children's Hospital and Brigham and Women's CF Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine (St. Louis), St Louis, Missouri
  - Rutgers Health, New Brunswick, New Jersey
  - New York Medical College (NYMC), Hawthorne, New York
  - Northwell LIJ Adult Cystic Fibrosis Center, New Hyde Park, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - University of Oklahoma Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University, Houston, Texas
  - University of Virginia Cystic Fibrosis Center, Charlottesville, Virginia